CLINICAL TRIAL: NCT02612142
Title: Efficacy of Exercise as an Adjunct Treatment for Clinically Depressed Inpatients During the Initial Stages of Antidepressant Therapy.
Brief Title: Physical EXercise as an Adjunct Treatment for Depression
Acronym: PEXAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Principal Investigator, Fabien Legrand, PhD, Université de Reims Champagne-Ardenne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPSMM-2011
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- aerobic exercise (AE) (Experimental): Intervention type: Behavioral. Intervention name: Aerobic exercise Intervention description: 10 days of daily aerobic exercise (brisk walking, jogging); duration: 30 minutes per session; intensity: 65%-75% of age-predicted maximal heart rate. All participants were treated with either paroxetine (20-50mg/day), fluoxetine (20-80mg/day) or bupropion (100-200mg/day).
  Interventions: Behavioral: physical exercise
- stretching exercise (ST) (Sham Comparator): Intervention type: Behavioral. Intervention name: Stretching exercise Intervention description: 10 days of daily stretching exercise; duration: 30 minutes per session. All participants were treated with either paroxetine (20-50mg/day), fluoxetine (20-80mg/day) or bupropion (100-200mg/day).
  Interventions: Behavioral: physical exercise
- no intervention (NI) (No Intervention): No behavioral intervention. All participants were treated with either paroxetine (20-50mg/day), fluoxetine (20-80mg/day) or bupropion (100-200mg/day).

INTERVENTIONS:
Behavioral: physical exercise — endurance-training or stretching (sham exercise)
  Arms: aerobic exercise (AE); stretching exercise (ST)

SUMMARY:
35 participants diagnosed with major depressive disorder were randomized in 3 intervention groups: (1) aerobic exercise (AE) ; (2) placebo (stretching) exercise (ST); and (3) no intervention (control group; NI). The intervention length was 10 consecutive days. In groups 1 (aerobic exercise) and 2 (sham exercise), participants exercised for 30 minutes each day. Depressive symptoms were assessed the day before the beginning of intervention and the day after the end of intervention for participants of both groups.

DETAILED DESCRIPTION:
In the aerobic exercise (AE) group, the intervention consisted of 30 minutes of daily brisk walking or jogging. This was done individually and supervised. Participants who missed > 2 training sessions were considered as non-completers. Exercise intensity had to be maintained within 65%-75% of age-predicted maximal heart rate, as commonly prescribed in studies using aerobic exercise to alleviate depression. Heart rate monitoring devices were used.

Participants in the stretching (ST) group also performed a daily 30 minutes exercise program but this was "sham" exercise, consisting of stretching exercises. Several muscle groups (thighs, calves, gluteal, shoulders, back) were stretched for 60 seconds, with equivalent resting intervals between stretching series. These activities were also individual and supervised. As was the case for the AE intervention, participants who missed > 2 training sessions were considered as non-completers.

Participants in the control (NI) group received no intervention other than prescribed medication.

All participants started antidepressants within less than 2 weeks before study entry.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of major depressive disorder (MDD)
* antidepressant drug therapy initiated for less than 2 weeks
* score of 29 or more on the Beck depression inventory

Exclusion Criteria:

* medical contraindication for exercise practice
* inability to understand written French
* beta-blocking drugs or another forms of antidepressant therapy (sleep deprivation, electroconvulsive therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Score change on the 21-item Beck depression inventory (BDI-II). Each item has a set of severity-graded self-evaluative statements that are rated 0 (neutral) to 3 (maximum severity). | Baseline and 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Zodi Imad, MD, Principal Investigator — Etablissement Public de Santé Mentale de la Marne